CLINICAL TRIAL: NCT02840643
Title: Combined Constraint Therapy and Bimanual Therapy for Children With Unilateral Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIMT-HABIT
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Hemiplegia; Cerebral Palsy
Keywords: hemispherectomy; brain; hand function
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Constraint Therapy and Bimanual Therapy (Experimental): Children in this arm will receive 90 hours (6 hrs/day, 5 days/week, 3 weeks) of Intensive Hand Therapy (constraint therapy), followed by 90 hours (6 hrs/day, 5 days/week, 3 weeks) of Intensive Bimanual Hand Therapy (bimanual therapy). During constraint therapy, children will wear a mitt over their less-impaired hand and actively use their more-impaired hand in therapy. Therapy will involve playing games, practicing activities of daily living, doing arts and crafts, and practicing repetitive hand movements. During bimanual therapy, children will actively use both hand in therapy. Therapy will involve playing games, practicing activities of daily living, doing arts and crafts, and practicing repetitive hand movements.
  Interventions: Behavioral: Bimanual hand therapy; Behavioral: Constraint therapy
- Bimanual Therapy and Constraint Therapy (Experimental): Children in this arm will receive 90 hours (6 hrs/day, 5 days/week, 3 weeks) of Intensive Bimanual Hand Therapy (bimanual therapy), followed by 90 hours (6 hrs/day, 5 days/week, 3 weeks) of Intensive Hand Therapy (constraint therapy). During bimanual therapy, children will actively use both hand in therapy. Therapy will involve playing games, practicing activities of daily living, doing arts and crafts, and practicing repetitive hand movements. During constraint therapy, children will wear a mitt over their less-impaired hand and actively use their more-impaired hand in therapy. Therapy will involve playing games, practicing activities of daily living, doing arts and crafts, and practicing repetitive hand movements.
  Interventions: Behavioral: Bimanual hand therapy; Behavioral: Constraint therapy

INTERVENTIONS:
Behavioral: Bimanual hand therapy — Children will receive 90 hours (6 hrs/day, 5 days/week, 3 weeks) of intensive bimanual hand therapy, which involves actively using both hands in play-based activities, games, arts and crafts, and activities of daily living. The different arms of the study will receive blocks of unimanual (constraint) therapy and bimanual therapy, in different orders.
Behavioral: Constraint therapy — Children will receive 90 hours (6 hrs/day, 5 days/week, 3 weeks) of intensive constraint therapy, which involves actively using the impaired hand in play-based activities, games, arts and crafts, and activities of daily living. The different arms of the study will receive blocks of unimanual (constraint) therapy and bimanual therapy, in different orders.

SUMMARY:
To examine efficacy of combined unimanual and bimanual intensive therapy in children with unilateral brain injury. A key question in hemiplegia therapy is whether the affected hand should be trained alone or in tandem with the other hand. In constraint-induced movement therapy (CIMT), a participant's less-affected upper extremity is restricted with a sling, cast, or mitt, while the participant actively uses the affected arm and hand in skill-based therapeutic activities. Bimanual therapy, in contrast, engages both hands in therapeutic movement. Since constraint and bimanual therapy target different aspects of hand use, they could have synergistic effects on hand function when given in combination.

DETAILED DESCRIPTION:
Children with hemiplegia will be given an intensive hand therapy protocol for six weeks (6 hrs/day, 5 days/week - total of 180 hours. Therapy will be given in two blocks.

In one block (3 weeks, 90 hours of therapy), children will receive constraint-induced movement therapy (CIMT), also known as constraint therapy. During CIMT, children wear a mitt over their less-affected hand, which restricts use of that hand. Children engage in intensive therapy to improve active range of motion, strength, motor control and sensory awareness of the affected hand. Activities are functional and play based. Daily structure of therapy includes: morning gym, fine motor, gross motor, sensory motor, therapeutic feeding, sports and self care activities. During training, children perform play-based and functional activities with the affected hand. Example activities include playing card and board games, arts and crafts, and activities that provide sensory stimulation to the affected hand, such as finger painting. Activities also include stretching and strengthening exercises.

In one block (3 weeks, 90 hours of therapy), children will receive bimanual therapy. During bimanual therapy, children do not wear a mitt over the less-affected hand. Children will be provided individualized activities that facilitated active use of both hands. Therapists will adapt and grade activities and guided children to problem solve for success. Bimanual activities include self-care (tying shoes, zippering, cutting food), sports activities, and manipulation of classroom tools (cutting with scissors).

Before the intervention begins, children will be randomized to one of two arms. In Arm 1, children will receive 3 weeks of CIMT followed by 3 weeks of bimanual therapy. In Arm 2, children will receive 3 weeks of bimanual therapy followed by 3 weeks of CIMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegia.
* Wrist range of motion of at least 10 degrees.
* Able to follow directions.
* Experience attending day programs without the child's home caregiver present (i.e. school, daycare).

Exclusion Criteria:

* Uncorrected vision problems.
* Inability to communicate or follow directions.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2011-07; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment after therapy | Day 1 of Intervention and day 180 of intervention
  The Assisting Hand Assessment (AHA) measures how well children use both hands in bimanual activities.

SECONDARY OUTCOMES:
Change in Assisting Hand Assessment after therapy follow-up | Day 1 of Intervention and two months after last day of intervention
  The Assisting Hand Assessment (AHA) measures how well children use both hands in bimanual activities.
Change in Assisting Hand Assessment after each three-week block of therapy | Day 1 of Intervention, end of third week of intervention, and end of sixth week of intervention
  The Assisting Hand Assessment (AHA) measures how well children use both hands in bimanual activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Blythedale Children's Hospital, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided